CLINICAL TRIAL: NCT06675513
Title: A Clinical Study on the Safety and Efficacy of GCC Targeting CAR-T Cells (WD-01) for Metastatic Colorectal Cancer
Brief Title: Autologous CAR-T Cells (WD-01) for Metastatic Colorectal Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wondercel Biotech (ShenZhen) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-GCC-WD-01
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: CRC (Colorectal Cancer); Metastatic Colorectal Cancer
Keywords: Autologous CAR-T therapy; WD-01; Wondercel
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single dose injection of WD-01 (Experimental): Dose escalation will be performed for the single dose injection of WD-01 for treating mCRC
  Interventions: Biological: An armored GCC targeting WD-01 CAR-T to treat cancer patients Other Name:

INTERVENTIONS:
Biological: An armored GCC targeting WD-01 CAR-T to treat cancer patients Other Name: — Autologous WD-01 CAR-T therapy with Wondercel's "Warrior" armor strategy will be explored for its advantage over other armor platforms.

SUMMARY:
This is an investigator initiated trial to assess the efficacy and safety of a GCC-targeting CAR-T therapy (WD-01) in the metastatic colorectal cancer.

DETAILED DESCRIPTION:
The study will use autologous T cells collected from enrolled patient, modified using a 2nd generation CAR bearing lentiviral vector, to treat metastatic colorectal cancer patients. The antigen-binding site of the CAR molecule recognizes GCC as the target.

The main questions it aims to answer are: • What is the maximum tolerated dose (MTD) of GCC-CAR-T therapy in the autologous CAR-T cell treatments? • What are the dose-limiting toxicities (DLT) and treatment-emergent adverse events (TEAE)? • What is the treatment efficacy, as measured by objective response rate (ORR) and progression-free survival (PFS)? Investigators will assess whether the WD-01 CAR-T cells have good safety and efficacy in treating colorectal cancer. Participants will receive WD-01 GCC-CAR-T cells through a 3+3 dose escalation scheme. • Undergo chemotherapy pre-conditioning before CAR-T infusion. • Be monitored for adverse events, immune response, and disease progression.

The study will collect data on both short-term outcomes (within the first few months post-treatment) and long-term safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed colorectal cancer. Immunohistochemistry (IHC) assessment shows GCC expression in tumor lesions of ≥1+ in an average of over 40% of the area (evaluated by randomly selecting at least five tumor regions).

Patients with metastatic colorectal cancer who have failed second-line treatment.

At least one measurable extracranial lesion per RECIST version 1.1 criteria. Expected survival of ≥90 days.

Normal function of major organs, meeting the following criteria:

1. ECOG performance status of 0-1 or KPS score >70.
2. Hematology parameters meeting: Hemoglobin (HB) ≥80 g/L, Absolute Neutrophil Count (ANC) ≥1.5 × 10^9/L, Platelets (PLT) ≥80 × 10^9/L, Lymphocytes (LY) ≥0.5 × 10^9/L.
3. Biochemistry parameters meeting: Total Bilirubin (TBIL) ≤2.0 × ULN (upper limit of normal); ALT and AST ≤2.5 × ULN; Serum Creatinine (Cr) ≤1 × ULN, Creatinine Clearance Rate >40 mL/min (by Cockcroft-Gault formula).
4. Left ventricular ejection fraction >55%. Women of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days prior to enrollment and agree to use appropriate contraception during the study and for 8 weeks after the last CAR-T administration (women who have undergone sterilization or have been postmenopausal for at least 2 years are considered not of childbearing potential).

Voluntary participation in the study, with signed informed consent, good compliance, and willingness to cooperate with follow-up.

Exclusion Criteria:

* Pregnant or lactating women. Receipt of small molecule chemotherapy, targeted agents, other investigational drugs, or monoclonal antibodies within 14 days prior to cell collection for enrollment.

Participation in other clinical trials within 4 weeks prior to the start of this study.

Uncontrolled hypertension that cannot be adequately managed with a single antihypertensive drug (systolic BP >160 mmHg, diastolic BP >100 mmHg), myocardial ischemia or infarction of grade ≥1, arrhythmia of grade ≥1 (including QT interval ≥440 ms), or cardiac insufficiency.

Long-standing, unhealed wounds or fractures. History of substance abuse that cannot be discontinued or a history of psychiatric disorders.

Severe intestinal adhesions, bowel obstruction, or conditions that may cause bowel perforation or abdominal wall fistula after treatment.

Uncontrolled or active fungal, bacterial, viral, or other infections. Grade ≥2 hematologic toxicity or grade ≥3 non-hematologic toxicity at enrollment as per NCI-CTCAE version 5.0 criteria.

Known HIV infection or active hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive) infection.

Presence of indwelling catheters or drainage tubes (e.g., biliary drainage tubes or thoracic/abdominal drainage tubes or pericardial catheters). Use of specialized central venous catheters is permitted.

Severe malnutrition (for patients <70 years, BMI <18.5 kg/m^2; for patients ≥70 years, BMI <20 kg/m^2).

History of severe allergic reactions to key therapeutic agents in this study (including fludarabine, cyclophosphamide, mesna, tocilizumab, and anti-infective drugs used during preconditioning).

History of disseminated intravascular coagulation (DIC), deep vein thrombosis, or pulmonary embolism within 6 months prior to enrollment.

History of autoimmune diseases that cause terminal organ damage or require systemic immunosuppressive/systemic disease-modifying drugs within 2 years prior to enrollment (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus).

Any disease that may interfere with the safety or efficacy assessment of the study treatment.

Female participants who are unwilling to use contraception from the time of consent until 6 months after completing CAR-T cell infusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-18 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Within the first month post-infusion
  The highest dose of GCC-CAR-T cells that can be administered without causing unacceptable side effects, measured during the dose escalation phase.
Dose-Limiting Toxicities (DLT) | Within the first month post-infusion
  The incidence of treatment-related toxicities that prevent further dose escalation.
Treatment-Emergent Adverse Events (TEAE) | From the administration of WD-01 CAR-T cells through six months post-infusion
  The frequency and severity of adverse events that arise following the administration of WD-01 CAR-T cells.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Measured between 1 and 6 months after treatment
  The proportion of patients with a measurable reduction in tumor size (complete or partial response) following GCC-CAR-T therapy.
Progression-Free Survival (PFS) | From the start of treatment up to 5 years
  The length of time during and after treatment that the patient lives without disease progression.
Overall Survival (OS) | From the start of treatment up to maximum follow-up period of five years
  The duration from the start of treatment to the time of death from any cause.
Duration of Response (DOR) | From the administration of WD-01 CAR-T cells to a maximum follow-up period of five years
  The time from initial tumor response (CR or PR) to disease progression or relapse or any cause of death.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Huazhong University of Science and Technology Union Hospital (Nanshan Hospital), Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No